CLINICAL TRIAL: NCT06900062
Title: The C-BRIDGE Study: China Bronchiectasis Research Involving Databases, Genomics, and Endotyping
Status: Recruiting | Type: Observational
Sponsor: Shanghai Pulmonary Hospital, Shanghai, China (Other)
Responsible Party: Principal Investigator, Gao Yong-hua, Associate Professor, Shanghai Pulmonary Hospital, Shanghai, China
Other Study IDs: 2024ZD0529700
Record Dates: First submitted 2025-03-23; First posted 2025-03-28 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-04

CONDITIONS: Bronchiectasis Adult
Keywords: bronchiectasis; phenotype; endotype; multi-omics; precision medicine
MeSH Terms: conditions — Bronchiectasis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 1. Whole blood, DNA, and plasma
  2. Sputum and sputum supernatant
  3. Bronchoalveolar lavage fluid (BALF); Bronchial epithelium collected via bronchoscopy
  4. Nasal swabs and nasal lavage fluid
  5. Urine
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients with bronchiectasis: Adult patients diagnosed with bronchiectasis who meet the study's inclusion criteria

SUMMARY:
Bronchiectasis is a heterogeneous airway disease with diverse causes, making precise diagnosis, prognosis, and treatment response prediction challenging. Identifying patient subgroups (phenotypes) and molecular profiles (endotypes) can enhance individualized assessment and management. While prior studies, primarily in European populations, have identified key phenotypes and endotypes, their relevance to Chinese patients remains unclear due to geographic and clinical differences. Specific causes of bronchiectasis, such as allergic bronchopulmonary aspergillosis (ABPA) and primary ciliary dyskinesia (PCD), may also exhibit distinct pathophysiology requiring further exploration. The C-BRIDGE Study seeks to characterize phenotypes and endotypes in Chinese bronchiectasis patients during stable disease and exacerbations, evaluate differences in clinical outcomes across these subgroups, and develop personalized medicine strategies based on these findings, applicable in China and globally.

Primary Objective: To identify molecular endotypes of bronchiectasis that accurately predict prognosis and guide treatment responses.

Secondary Objectives:

To characterize molecular endotypes of stable bronchiectasis in Chinese patients.

To define molecular endotypes of bronchiectasis exacerbations in Chinese patients.

To investigate molecular endotypes specific to allergic bronchopulmonary aspergillosis (ABPA).

To explore genotypes and inflammatory endotypes of cystic fibrosis (CF) and primary ciliary dyskinesia (PCD) in Chinese patients.

To validate candidate biomarkers for stable and exacerbation endotypes to support stratified medicine.

To conduct in vivo or in vitro proof-of-concept studies using phenotypic data to identify patient subgroups likely to benefit from specific pharmacological interventions.

Study Design: This observational cohort study will link identified patient subgroups with meaningful clinical outcomes to inform prognosis and optimize treatment strategies.

DETAILED DESCRIPTION:
Bronchiectasis is a common, heterogeneous chronic airway disease that remains understudied in clinical and translational research. Although several phenotypes and endotypes have been identified-primarily in European populations-data from Chinese patients are limited. Racial and geographic differences suggest that bronchiectasis phenotypes and endotypes in China may differ from those in Western cohorts. Recent controlled trials have failed to meet primary endpoints, likely due to insufficient identification of patient subgroups that optimally respond to antibiotics, mucoactive agents, or anti-inflammatory therapies. The C-BRIDGE Study seeks to address this gap by exploring the clinical, genomic, microbiological, inflammatory, and functional heterogeneity of bronchiectasis in Chinese patients to define molecular endotypes for stratified assessment and management.

Study Aims and Objectives:

1. Characterize molecular endotypes of stable bronchiectasis in Chinese patients.
2. Identify molecular endotypes of bronchiectasis exacerbations in Chinese patients.
3. Investigate molecular endotypes in patients with allergic bronchopulmonary aspergillosis (ABPA).
4. Develop a screening algorithm and elucidate genotypes and inflammatory endotypes of cystic fibrosis (CF) and primary ciliary dyskinesia (PCD) in China.
5. Validate candidate biomarkers for stable and exacerbation endotypes to enable stratified medicine.
6. Perform in vivo and in vitro proof-of-concept studies using phenotypic data to pinpoint patient subgroups likely to benefit from specific pharmacological treatments.

Study Design:

Observational cohort study.

Study Methods:

A target of 1,500 patients with bronchiectasis will be recruited across participating centers for an observational study with the following aims:

Aim 1: Stable Disease Endotyping Up to 1,500 patients will be studied to define and validate endotypes of stable bronchiectasis. Data collection will include clinical assessments, sputum and nasal microbiome analysis, sputum proteomics, nasal and airway transcriptomics, single-cell sequencing of bronchoalveolar lavage fluid (BALF), and measurement of inflammatory markers in systemic, nasal, sputum, and BALF samples. A sub-study (n=100) will use air-liquid interface cultures of primary airway epithelial cells to assess responses to various stimuli and pharmacological interventions.

Aim 2: Exacerbation Endotyping A subset of 200 patients will be evaluated during exacerbations to replicate the phenotyping approach. This will involve analyzing changes from baseline in microbiome, proteomics, metabolomics, and other markers to identify clusters linked to exacerbation onset, progression, and outcomes.

Aim 3: Allergic Bronchopulmonary Aspergillosis (ABPA) Subgroup Analysis A subset of 150 patients with ABPA will be studied to investigate molecular endotypes by integrating single-cell sequencing, microbiome, mycobiome, proteomics, metabolomics, and other markers to identify clusters associated with exacerbation, recurrence, and treatment responses.

Aim 4: Idiopathic Bronchiectasis and Genetic Screening Patients with idiopathic bronchiectasis will be screened for cystic fibrosis, CFTR-related disorders, and primary ciliary dyskinesia (PCD) to identify genotypes and inflammatory endotypes. This will integrate genomics, microbiome, proteomics, and metabolomics to explore associations among phenotypes, genotypes, endotypes, and prognosis.

Aim 5: Biomarker Validation and Prediction Model Development Candidate phenotypes and endotypes will be externally validated using registered, ethically approved biobanks. Validated biomarkers will be correlated with clinically meaningful outcomes, such as treatment responses, to enable their use in stratified medicine. Clinical data and validated biomarkers will be integrated to construct and validate prediction models for exacerbation frequency, time to first exacerbation, and lung function decline.

Participants will visit the Clinical Research Centre at least once for sampling and clinical data collection, with consent obtained to link their samples to the C-BRIDGE database.

Ethics Approval:

Approved by the Ethics Committee of Shanghai Pulmonary Hospital and other participating centers.

Expected Outcomes:

The C-BRIDGE Study will establish detailed molecular endotypes of bronchiectasis in Chinese patients, facilitating precise prognosis prediction and tailored treatment strategies. By identifying and validating patient subgroups and biomarkers, it will provide a foundation for personalized medicine in bronchiectasis management, with potential relevance in China and worldwide.

ELIGIBILITY:
Inclusion Criteria:

* A prior CT scan confirming bronchiectasis, accompanied by a compatible clinical syndrome including cough, sputum production, and/or recurrent respiratory tract infections.
* At the screening visit, participants must have been clinically stable for 4 weeks, defined as no antibiotic or corticosteroid treatment for a pulmonary exacerbation in the preceding 4 weeks.

Exclusion Criteria:

* Inability to provide informed consent
* Age under 18 years
* Patients with active tuberculosis
* Use of antibiotics or corticosteroids for a pulmonary exacerbation within the past 4 weeks

Ages: 18 Years to 85 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients with bronchiectasis
Sampling Method: Non-Probability Sample
Enrollment: 1500 (Estimated)
Dates: Start 2025-04-06 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2029-01-31 (Estimated)

PRIMARY OUTCOMES:
Frequency of bronchiectasis exacerbations | 2 years
  Worsening of respiratory symptoms, as defined by the EMBARC/BRR criteria (Eur Respir J. 2017;49(6):1700051), requiring adjustments to treatment strategies.

SECONDARY OUTCOMES:
Time to the first exacerbation | 2 years
  Worsening of respiratory symptoms, as defined by the EMBARC/BRR criteria (Eur Respir J. 2017;49(6):1700051), requiring adjustments to treatment strategies.
The Quality of Life Bronchiectasis Respiratory Symptom Scales (QOL-B-RSS) | 2 years
  The Quality-of-Life-Bronchiectasis (QoL-B) questionnaire is a disease-specific survey designed for patients with bronchiectasis. The Respiratory Symptoms scale is a component of the QoL-B questionnaire, with a scale range from 0 to 100. Higher scores on this scale signify a better health status. In bronchiectasis, the established minimal clinically important difference (MCID) is 8 points.
The Bronchiectasis Health Questionnaire (BHQ) | 2 years
  The BHQ is a brief, self-administered tool consisting of 10 items that assess health status over the previous 14 days. It uses 7-point Likert scales, with scores ranging from 0 to 100, where higher scores reflect better health-related quality of life (HRQoL). In bronchiectasis, the established minimal clinically important difference (MCID) is 3 points.
The Bronchiectasis Impact Measure (BIM) | 2 years
  The Bronchiectasis Impact Measure (BIM) is a validated patient-reported outcome measure for patients with bronchiectasis. The BIM includes eight domains (cough, sputum, breathlessness, tiredness, activity, general health, control, exacerbations) and is numbered 0-10. Higher scores on this scale signify a greater impact of these domains on daily life. In bronchiectasis, the minimal clinically important difference (MCID) for each domain as 1.5 points on a 10-point scale.
The St Georges Respiratory Questionnaire (SGRQ) | 2 years
  St.George Respiratory Questionnaire (SGRQ): a validated questionnaire for use in bronchiectasis population. This questionnaire is structured into 3 main components: symptoms, activity and impacts.
  Scale range is 0-100, where lower scores correspond to the better health status.
  Each questionnaire response has a unique empirically derived "weight".
  Each component of the questionnaire is scored separately in three steps:
  i. The weights for all items with a positive responses are summed. ii. The weights for missed items are deducted from the maximum possible weight for each component. The weights for all missed items are deducted from the maximum possible weight for the Total score.
  iii. The score is calculated by dividing the summed weights by the adjusted maximum possible weight for that component and expressing the result as a percentage The Total score is calculated in similar way. In bronchiectasis, the established MCID is 4 points.
The bronchiectasis exacerbation and symptom tool (BEST) | 2 years
  The Bronchiectasis Exacerbation and Symptom Tool (BEST) is a validated questionnaire designed to evaluate daily symptoms in patients with bronchiectasis. It has a maximum score of 26, with higher scores reflecting a greater symptom burden. In bronchiectasis, the minimal clinically important difference (MCID) is 4 points.
Bronchiectasis Symptom VAS (BS-VAS) | 2 years
  The Bronchiectasis Symptom Visual Analogue Scale (BS-VAS) is a simple, patient-reported tool designed to quantify the severity of individual symptom burden in patients with bronchiectasis. It consists of 11 separate 100-mm horizontal visual analogue scales, each assessing a different core symptom: cough, sputum volume, sputum colour, sputum viscosity, dyspnoea, fatigue, wheezing, chest tightness, chest pain, exercise tolerance, and haemoptysis.
  Patients are instructed to mark a vertical line on each 10-mm scale to indicate symptom severity over the past 24 hours, with the left anchor (0 mm) defined as "No symptom at all" and the right anchor (10 mm) defined as "Worst imaginable". Each item is measured from 0 to 10 mm (scored 0-10 with one decimal place).
Forced expiratory volume in 1 second (FEV1) | 2 years
  Spirometry
Hospitalization for severe exacerbations | 2 years
  Admission to hospital for an exacerbation meeting the EMBARC/BRR exacerbation
All cause mortality | 3 years
  Survival during the study

CONTACTS AND LOCATIONS:
Overall Officials: Yong-hua Gao, Ph.D., Principal Investigator — Shanghai Pulmonary Hospital, Shanghai, China
Locations (9):
- China (9):
  - Lin Liu, Guiyang, Guizhou
  - Lei Song, Changchun, Jilin
  - Qian Qi, Jinan, Shangdong
  - He-feng Chen, Shanghai, Shanghai Municipality
  - Zhou-fang Mei, Shanghai, Shanghai Municipality
  - Jun She, Shanghai, Shanghai Municipality
  - Xue-ling Wu, Shanghai, Shanghai Municipality
  - Yong-hua Gao, Shanghai, Shanghai Municipality
  - Xiao-long Ma, Jiaxing, Zhejiang

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gao Y, Richardson H, Dicker AJ, Barton A, Kuzmanova E, Shteinberg M, Perea L, Goeminne PC, Cant E, Hennayake C, Pollock J, Abo Leyah H, Choi H, Polverino E, Blasi F, Welte T, Aliberti S, Long M, Shoemark A, Sibila O, Huang JTJ, Chalmers JD. Endotypes of Exacerbation in Bronchiectasis: An Observational Cohort Study. Am J Respir Crit Care Med. 2024 Jul 1;210(1):77-86. doi: 10.1164/rccm.202310-1729OC. PMID 38717347
- [Background] Choi H, Ryu S, Keir HR, Giam YH, Dicker AJ, Perea L, Richardson H, Huang JTJ, Cant E, Blasi F, Pollock J, Shteinberg M, Finch S, Aliberti S, Sibila O, Shoemark A, Chalmers JD. Inflammatory Molecular Endotypes in Bronchiectasis: A European Multicenter Cohort Study. Am J Respir Crit Care Med. 2023 Dec 1;208(11):1166-1176. doi: 10.1164/rccm.202303-0499OC. PMID 37769155
- [Background] Shoemark A, Shteinberg M, De Soyza A, Haworth CS, Richardson H, Gao Y, Perea L, Dicker AJ, Goeminne PC, Cant E, Polverino E, Altenburg J, Keir HR, Loebinger MR, Blasi F, Welte T, Sibila O, Aliberti S, Chalmers JD. Characterization of Eosinophilic Bronchiectasis: A European Multicohort Study. Am J Respir Crit Care Med. 2022 Apr 15;205(8):894-902. doi: 10.1164/rccm.202108-1889OC. PMID 35050830
- [Background] Chalmers JD, Aliberti S, Filonenko A, Shteinberg M, Goeminne PC, Hill AT, Fardon TC, Obradovic D, Gerlinger C, Sotgiu G, Operschall E, Rutherford RM, Dimakou K, Polverino E, De Soyza A, McDonnell MJ. Characterization of the "Frequent Exacerbator Phenotype" in Bronchiectasis. Am J Respir Crit Care Med. 2018 Jun 1;197(11):1410-1420. doi: 10.1164/rccm.201711-2202OC. PMID 29357265
- [Background] Huang JT, Cant E, Keir HR, Barton AK, Kuzmanova E, Shuttleworth M, Pollock J, Finch S, Polverino E, Bottier M, Dicker AJ, Shoemark A, Chalmers JD. Endotyping Chronic Obstructive Pulmonary Disease, Bronchiectasis, and the "Chronic Obstructive Pulmonary Disease-Bronchiectasis Association". Am J Respir Crit Care Med. 2022 Aug 15;206(4):417-426. doi: 10.1164/rccm.202108-1943OC. PMID 35436182
- [Background] Shoemark A, Griffin H, Wheway G, Hogg C, Lucas JS; Genomics England Research Consortium; Camps C, Taylor J, Carroll M, Loebinger MR, Chalmers JD, Morris-Rosendahl D, Mitchison HM, De Soyza A; Genomics England Research Consortium:; Brown D, Ambrose JC, Arumugam P, Bevers R, Bleda M, Boardman-Pretty F, Boustred CR, Brittain H, Caulfield MJ, Chan GC, Fowler T, Giess A, Hamblin A, Henderson S, Hubbard TJP, Jackson R, Jones LJ, Kasperaviciute D, Kayikci M, Kousathanas A, Lahnstein L, Leigh SEA, Leong IUS, Lopez FJ, Maleady-Crowe F, McEntagart M, Minneci F, Moutsianas L, Mueller M, Murugaesu N, Need AC, O'Donovan P, Odhams CA, Patch C, Perez-Gil D, Pereira MB, Pullinger J, Rahim T, Rendon A, Rogers T, Savage K, Sawant K, Scott RH, Siddiq A, Sieghart A, Smith SC, Sosinsky A, Stuckey A, Tanguy M, Taylor Tavares AL, Thomas ERA, Thompson SR, Tucci A, Welland MJ, Williams E, Witkowska K, Wood SM. Genome sequencing reveals underdiagnosis of primary ciliary dyskinesia in bronchiectasis. Eur Respir J. 2022 Nov 17;60(5):2200176. doi: 10.1183/13993003.00176-2022. Print 2022 Nov. PMID 35728977
- [Background] Hill AT, Haworth CS, Aliberti S, Barker A, Blasi F, Boersma W, Chalmers JD, De Soyza A, Dimakou K, Elborn JS, Feldman C, Flume P, Goeminne PC, Loebinger MR, Menendez R, Morgan L, Murris M, Polverino E, Quittner A, Ringshausen FC, Tino G, Torres A, Vendrell M, Welte T, Wilson R, Wong C, O'Donnell A, Aksamit T; EMBARC/BRR definitions working group. Pulmonary exacerbation in adults with bronchiectasis: a consensus definition for clinical research. Eur Respir J. 2017 Jun 8;49(6):1700051. doi: 10.1183/13993003.00051-2017. Print 2017 Jun. PMID 28596426
- [Background] Aliberti S, Lonni S, Dore S, McDonnell MJ, Goeminne PC, Dimakou K, Fardon TC, Rutherford R, Pesci A, Restrepo MI, Sotgiu G, Chalmers JD. Clinical phenotypes in adult patients with bronchiectasis. Eur Respir J. 2016 Apr;47(4):1113-22. doi: 10.1183/13993003.01899-2015. Epub 2016 Feb 4. PMID 26846833
- [Background] Chalmers JD, Aliberti S, Polverino E, Vendrell M, Crichton M, Loebinger M, Dimakou K, Clifton I, van der Eerden M, Rohde G, Murris-Espin M, Masefield S, Gerada E, Shteinberg M, Ringshausen F, Haworth C, Boersma W, Rademacher J, Hill AT, Aksamit T, O'Donnell A, Morgan L, Milenkovic B, Tramma L, Neves J, Menendez R, Paggiaro P, Botnaru V, Skrgat S, Wilson R, Goeminne P, De Soyza A, Welte T, Torres A, Elborn JS, Blasi F. The EMBARC European Bronchiectasis Registry: protocol for an international observational study. ERJ Open Res. 2016 Jan 20;2(1):00081-2015. doi: 10.1183/23120541.00081-2015. eCollection 2016 Jan. PMID 27730179